CLINICAL TRIAL: NCT02962635
Title: A Pilot stuDy to Investigate the Role of Biomarkers and Bioimpedance technologY to Assess VolumE Status In Patients underGoing Hemodialysis Treatment
Brief Title: Role of Biomarkers in Patients Undergoing Dialysis Treatment
Acronym: DRYWEIGHT
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: DRYWEIGHT
Record Dates: First submitted 2016-11-02; First posted 2016-11-11 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Volemia in Dialysis Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis patients: A total of 30 patients
  - measuring volume status by bioelectrical impedance measurement as well as clinical evaluation and comparing with the novel biomarker
  Interventions: Device: bioelectrical impedance measurement and biomarker measurement
- Peritoneal dialysis patients: A total of 15 patients
  - measuring volume status by bioelectrical impedance measurement as well as clinical evaluation and comparing with the novel biomarker
  Interventions: Device: bioelectrical impedance measurement and biomarker measurement

INTERVENTIONS:
Device: bioelectrical impedance measurement and biomarker measurement — Measuring volume status with bioelectrical impedance measurement and comparing with biomarker level

SUMMARY:
A precise volume status assessment is critical to improve outcome of patients on dialysis. Yet, accurate assessment of fluid status remains a challenge. Currently, this is performed by clinical evaluation and regular weight measurements before and after dialysis, which is not always accurate. Moreover, bioimpedance technology is used in some centers for quantitative assessment of total body water. This approach has been validated for the assessment of volume status in dialysis patients, but requires the acquisition of specific tools and is time consuming. So far, no biomarker has been validated to quantify volume status in dialysis patients. Application of biomarkers might contribute to a better dialysis prescription and therefore to outcome improvement in dialysis. The investigators aim to investigate the role of a novel biomarkers (sCD146) to assess volume status in dialysis patients

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patient on dialysis since > 1 month
* Voluntarily signed informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women and women who plan to get pregnant during study
* Incapability of following the study protocol
* Acute illness
* Hospitalizations in the last week before inclusion
* Cardiac pacemakers or defibrillators
* Limb amputation or other factors precluding a reliable bioimpedance measurement (unreliable bioimpedance measurement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage renal failure on hemodialysis and peritoneal dialysis
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-10; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Correlation of sCD146 level with overhydration assessed by bioimpedance technology | 3 weeks to 3 months
  For hemodialysis patients measurements will be concluded within 3 weeks, for peritoneal dialysis patients measures will be concluded within 3 months

SECONDARY OUTCOMES:
Correlation of sCD146 level measured after dialysis and ultrafiltration rate | 3 weeks
  for hemodialysis patients measurements will be concluded within 3 weeks
Correlation of sCD146 level and clinical evaluation of volume status | 3 weeks to 3 months
  For hemodialysis patients measurements will be concluded within 3 weeks, for peritoneal dialysis patients measures will be concluded within 3 months
Correlation of sCD146 level and level of NT-proBNP | 3 weeks to 3 months
  For hemodialysis patients measurements will be concluded within 3 weeks, for peritoneal dialysis patients measures will be concluded within 3 months
Correlation of sCD146 level and mortality as assessed prospectively in 6 months follow-up | 6 months
Correlation of sCD146 level and hospitalizations as assessed prospectively in 6 months follow-up | 6 months
Correlation of sCD146 level and cardiovascular complications as assessed prospectively in 6 months follow-up | 6 months
Correlation of sCD146 level and shunt complications as assessed prospectively in 6 months follow-up | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Segerer, MD, Principal Investigator — University Hospital Zürich, Zürich, Switzerland
Locations (1):
- University Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided